CLINICAL TRIAL: NCT05024942
Title: Lung Ultrasound in Aortic Stenosis Patients Undergoing Transcatheter Aortic Valve Replacement: a Prospective Study
Brief Title: LUS in Aortic Stenosis Patients Undergoing TAVR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Francesca Graziani, MD (Unknown); Stefano Cangemi, MD (Unknown)
Responsible Party: Principal Investigator, Francesco Burzotta, MD, PhD, interventional cardiologist, Catholic University of the Sacred Heart
Other Study IDs: ID 3965
Record Dates: First submitted 2021-08-10; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Transcatheter Aortic Valve Replacement; Lung Ultrasound; Severe Aortic Valve Stenosis; Pulmonary Congestion
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Severe aortic stenosis patients undergoing TAVR: Severe aortic stenosis patients undergoing TAVR will be stratified according to LUS evaluated pulmonary congestion before and after TAVR
  Interventions: Procedure: Transfemoral TAVR (Transcatheter aortic valve replacement)

INTERVENTIONS:
Procedure: Transfemoral TAVR (Transcatheter aortic valve replacement) — Transfemoral transcatheter aortic valve replacement (TAVR) is a minimally invasive heart procedure to replace a narrowed aortic valve that fails to open properly (aortic valve stenosis) through an incision in the groin. All FDA approved transcatheter aortic prosthesys are allowed.

SUMMARY:
1. Introduction and aims:

   Transcatheter aortic valve replacement (TAVR) is the gold standard for the treatment of elderly patients with severe aortic valve stenosis (AS). AS causes left ventricular remodeling as well as left atrial enlargement, pulmonary artery and right ventricular changes, these changes, and whether they are reversible (reverse remodeling) are major determinants of outcome after TAVR. Heart Failure (HF) is the most frequent cause of cardiac re-hospitalization after TAVR. Most HF exacerbations are related to a progressive rise in cardiac filling pressures that precipitates pulmonary congestion and symptomatic decompensation. Traditionally, pulmonary congestion has been assessed by physical examination and chest radiography but clinical signs and symptoms of congestion are poor surrogates for ventricular filling pressures and are not reliable predictors of imminent hospitalization. Recently, lung ultrasonography (LUS) has been identified as a sensitive and semi-quantitative tool for the assessment of pulmonary congestion in HF. The technique is based on the detection of vertical echogenic artifacts arising from the pleural line, named "B-lines". The number of B-lines is associated with increased risk of adverse events during hospitalization and after hospital discharge. CLUSTER-HF Trial demonstrated that the routine incorporation of LUS during clinical follow-up of patients with recent acute decompensated HF without a surgically correctable cause, was associated with a risk reduction of adverse HF events, mainly urgent HF visits.

   Thus, LUS could represent a promising tool to detect pulmonary congestion related to AS. To date, there are no studies on the role of LUS in the context of AS and TAVR.

   The study hypothesis is that in patients with higher number of B-lines before-TAVR and after TAVR, the rate of adverse events during follow-up is higher.
2. Study design:

   This is a single center prospective study carried out at Fondazione Policlinico Gemelli IRCCS, Roma and involving patients with severe aortic stenosis submitted to TAVR treatment. The expected recruitment period is approximately one year For patients fulfilling inclusion/exclusion criteria, all data about clinical status leading to TAVR, exams and any specific documentation during hospitalization will be collected.
3. Number of patients:

   For the primary end-point, a sample-size of 91 is computed using the one-sample chi-square test and assuming a proportion of LUS-evaluated pulmonary congested patients before TAVR of 50% and a proportion of 35% of LUS-evaluated pulmonary congested patients after TAVR. To accommodate for possible missing investigations, sample size will be increased to 105 patients.

   The secondary end-point is the association between pre-TAVR and post-TAVR B-lines and long-term outcomes. Based on previous studies, the investigators know that the incidence of rehospitalization for heart failure during one-year after TAVR is 14% and that patients suffering from heart failure without LUS-evaluated pulmonary congestion are at very low risk of heart failure rehospitalization during follow-up. So, for sample size calculation of the secondary endpoint, the investigators estimated a cumulative incidence higher in the LUS- evaluated pulmonary congestion group with more than 16 B-lines on all scanning sites (30% of events during 1-year of follow-up) with a lower incidence of 8% in the remaining patients. With an HR of 5 favoring patients wit less than 15 B-Lines on all scanning, and aiming to a 2-sided alpha level of 0.05 and a power of 80% the investigators estimated 144 patients. To accommodate for possible missing investigations, sample size will be increased to 150 patients.
4. In-hospital study schedule:

   For each patient, the investigators will obtain from our general hospital database the following clinical data:
   * Demographic and clinical data documentation;
   * Clinical examination: before TAVR, before discharge and when adverse events occur;
   * Blood analysis;
   * TAVR procedural characteristics and complications.
5. Instrumental diagnostic exams (Echocardiography and lung ultrasound):

   Each patient will be evaluated before and after TAVR with a comprehensive echocardiogram and LUS for the evaluation of the pulmonary congestion. All the evaluations will be performed the day before TAVR and after TAVR.

   In consideration of the operator's dependence on ultrasound methods to reduce the error rate, all examinations will be performed by qualified personnel.
6. Clinical follow up assessment:

Clinical follow up information will be obtained from: visits, review of the patient's hospital record, personal communication with the patient's physician and review of the patient's chart, a telephone interview with the patient conducted by trained medical personnel The following information will be recorded: clinical status assessment, adverse event assessment, record cardiac medications.

ELIGIBILITY:
Inclusion Criteria:

* severe aortic stenosis,
* life expectancy >1 year,
* patient candidate to percutaneous transfemoral aortic valve implantation after formal indication of our "Heart Team".

Exclusion Criteria:

* clinical history of lung cancer or lung surgery, fibrothorax and pneumothorax, pulmonary fibrosis,
* patients undergoing urgent aortic valvuloplasty,
* patients admitted for cardiogenic shock,
* recent (within 1 month) pneumonia or ARDS (Acute Respiratory Distress Syndrome),
* lack of will to participate,
* more than moderate aortic regurgitation,
* valve-in-valve procedures,
* transapical and transaortic TAVR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing TAVR for severe aortic stenosis could participate in the study and therefore, be evaluated according to the selection criteria defined in the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
change of LUS-evaluated pulmonary congestion in patients with severe aortic stenosis undergoing TAVR | pre-intervention (baseline) and after the intervention within 72 hours

SECONDARY OUTCOMES:
to evaluate the possible prognostic role of LUS-evaluated pulmonary congestion at 12 months follow-up. | One year after hospital discharge.
  The main adverse events considered in the secondary end-point are: death from cardiovascular cause, hospitalization for HF and urgent medical visits for worsening dyspnea in the 12 months following discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico A. Gemelli. Università Cattolica del Sacro Cuore, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reardon MJ, Van Mieghem NM, Popma JJ, Kleiman NS, Sondergaard L, Mumtaz M, Adams DH, Deeb GM, Maini B, Gada H, Chetcuti S, Gleason T, Heiser J, Lange R, Merhi W, Oh JK, Olsen PS, Piazza N, Williams M, Windecker S, Yakubov SJ, Grube E, Makkar R, Lee JS, Conte J, Vang E, Nguyen H, Chang Y, Mugglin AS, Serruys PW, Kappetein AP; SURTAVI Investigators. Surgical or Transcatheter Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2017 Apr 6;376(14):1321-1331. doi: 10.1056/NEJMoa1700456. Epub 2017 Mar 17. PMID 28304219
- [Background] Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Feb 2;143(5):e35-e71. doi: 10.1161/CIR.0000000000000932. Epub 2020 Dec 17. PMID 33332149
- [Background] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053
- [Background] Treibel TA, Badiani S, Lloyd G, Moon JC. Multimodality Imaging Markers of Adverse Myocardial Remodeling in Aortic Stenosis. JACC Cardiovasc Imaging. 2019 Aug;12(8 Pt 1):1532-1548. doi: 10.1016/j.jcmg.2019.02.034. PMID 31395243
- [Background] Lindman BR, Stewart WJ, Pibarot P, Hahn RT, Otto CM, Xu K, Devereux RB, Weissman NJ, Enriquez-Sarano M, Szeto WY, Makkar R, Miller DC, Lerakis S, Kapadia S, Bowers B, Greason KL, McAndrew TC, Lei Y, Leon MB, Douglas PS. Early regression of severe left ventricular hypertrophy after transcatheter aortic valve replacement is associated with decreased hospitalizations. JACC Cardiovasc Interv. 2014 Jun;7(6):662-73. doi: 10.1016/j.jcin.2014.02.011. PMID 24947722
- [Background] Genereux P, Pibarot P, Redfors B, Mack MJ, Makkar RR, Jaber WA, Svensson LG, Kapadia S, Tuzcu EM, Thourani VH, Babaliaros V, Herrmann HC, Szeto WY, Cohen DJ, Lindman BR, McAndrew T, Alu MC, Douglas PS, Hahn RT, Kodali SK, Smith CR, Miller DC, Webb JG, Leon MB. Staging classification of aortic stenosis based on the extent of cardiac damage. Eur Heart J. 2017 Dec 1;38(45):3351-3358. doi: 10.1093/eurheartj/ehx381. PMID 29020232
- [Background] Vemulapalli S, Dai D, Hammill BG, Baron SJ, Cohen DJ, Mack MJ, Holmes DR Jr. Hospital Resource Utilization Before and After Transcatheter Aortic Valve Replacement: The STS/ACC TVT Registry. J Am Coll Cardiol. 2019 Mar 19;73(10):1135-1146. doi: 10.1016/j.jacc.2018.12.049. PMID 30871697
- [Background] Gheorghiade M, Follath F, Ponikowski P, Barsuk JH, Blair JE, Cleland JG, Dickstein K, Drazner MH, Fonarow GC, Jaarsma T, Jondeau G, Sendon JL, Mebazaa A, Metra M, Nieminen M, Pang PS, Seferovic P, Stevenson LW, van Veldhuisen DJ, Zannad F, Anker SD, Rhodes A, McMurray JJ, Filippatos G; European Society of Cardiology; European Society of Intensive Care Medicine. Assessing and grading congestion in acute heart failure: a scientific statement from the acute heart failure committee of the heart failure association of the European Society of Cardiology and endorsed by the European Society of Intensive Care Medicine. Eur J Heart Fail. 2010 May;12(5):423-33. doi: 10.1093/eurjhf/hfq045. Epub 2010 Mar 30. PMID 20354029
- [Background] Zile MR, Bennett TD, St John Sutton M, Cho YK, Adamson PB, Aaron MF, Aranda JM Jr, Abraham WT, Smart FW, Stevenson LW, Kueffer FJ, Bourge RC. Transition from chronic compensated to acute decompensated heart failure: pathophysiological insights obtained from continuous monitoring of intracardiac pressures. Circulation. 2008 Sep 30;118(14):1433-41. doi: 10.1161/CIRCULATIONAHA.108.783910. Epub 2008 Sep 15. PMID 18794390
- [Background] Rivas-Lasarte M, Maestro A, Fernandez-Martinez J, Lopez-Lopez L, Sole-Gonzalez E, Vives-Borras M, Montero S, Mesado N, Pirla MJ, Mirabet S, Fluvia P, Brossa V, Sionis A, Roig E, Cinca J, Alvarez-Garcia J. Prevalence and prognostic impact of subclinical pulmonary congestion at discharge in patients with acute heart failure. ESC Heart Fail. 2020 Oct;7(5):2621-2628. doi: 10.1002/ehf2.12842. Epub 2020 Jul 7. PMID 32633473
- [Background] Platz E, Campbell RT, Claggett B, Lewis EF, Groarke JD, Docherty KF, Lee MMY, Merz AA, Silverman M, Swamy V, Lindner M, Rivero J, Solomon SD, McMurray JJV. Lung Ultrasound in Acute Heart Failure: Prevalence of Pulmonary Congestion and Short- and Long-Term Outcomes. JACC Heart Fail. 2019 Oct;7(10):849-858. doi: 10.1016/j.jchf.2019.07.008. PMID 31582107
- [Background] Picano E, Scali MC, Ciampi Q, Lichtenstein D. Lung Ultrasound for the Cardiologist. JACC Cardiovasc Imaging. 2018 Nov;11(11):1692-1705. doi: 10.1016/j.jcmg.2018.06.023. PMID 30409330
- [Background] Araiza-Garaygordobil D, Gopar-Nieto R, Martinez-Amezcua P, Cabello-Lopez A, Alanis-Estrada G, Luna-Herbert A, Gonzalez-Pacheco H, Paredes-Paucar CP, Sierra-Lara MD, Briseno-De la Cruz JL, Rodriguez-Zanella H, Martinez-Rios MA, Arias-Mendoza A. A randomized controlled trial of lung ultrasound-guided therapy in heart failure (CLUSTER-HF study). Am Heart J. 2020 Sep;227:31-39. doi: 10.1016/j.ahj.2020.06.003. Epub 2020 Jun 15. PMID 32668323
- [Derived] Lillo R, Cangemi S, Graziani F, Locorotondo G, Pedicino D, Aurigemma C, Romagnoli E, Malara S, Meucci MC, Iannaccone G, Bianchini F, Nesta M, Bruno P, Lombardo A, Trani C, Burzotta F. Pulmonary congestion assessed by lung ultrasound in patients with severe aortic stenosis undergoing transcatheter aortic valve implantation: Prevalence and prognostic implications. Eur J Heart Fail. 2024 Oct;26(10):2107-2117. doi: 10.1002/ejhf.3365. Epub 2024 Jul 16. PMID 39014551